CLINICAL TRIAL: NCT01816555
Title: Vitamin D3 (Vit D3) Supplementation and T Cell Immunomodulation in Patients With Newly Diagnosed Operative Invasive Ductal Breast Carcinoma Stage I-II
Brief Title: Vitamin D3 (Vit D3) Supplementation and T Cell Immunomodulation in Patients With Newly Diagnosed Operative Invasive Ductal Breast Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to low accrual.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101813
Record Dates: First submitted 2013-02-06; First posted 2013-03-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2014-08

CONDITIONS: Newly Diagnosed Operative Invasive Ductal Breast Carcinoma Stage I-II
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D- Normal Level at Screening (Experimental): Subjects will have surgery as their initial breast therapy. If subjects have a normal level of Vitamin D(25-hydroxyVit D 30-100ng/mL), they will be assigned to this group.
  Interventions: Dietary Supplement: Vitamin D
- Vitamin D- Insufficient or Deficient Level at Screening (Experimental): Subjects will have surgery as their initial breast therapy. If subjects are insufficient (25-hydroxy Vit D 21-29 ng/mL)or deficient (25-hydroxyVit D <20ng/mL) Vitamin D levels, they will be assigned to this group.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Subjects will be assigned to a dosage level between 600IU daily and 10,000IU daily depending on their age, weight and current vitamin D level

SUMMARY:
This study is for adult females who have been newly diagnosed with breast cancer that includes surgery as part of standard cancer treatment. This is a research study combining Vitamin D (an over the counter medication) with the standard of care (or the established and approved treatment), surgery. Evidence shows that women who are Vitamin D3 deficient have a higher risk of breast cancer and breast cancer recurrence. The purpose of this study is to find out the effects of Vitamin D3 during the treatment period for Stage I-II breast cancer. Screening tests will be done to determine if subjects are eligible to participate in this study. If subjects are eligible and they agree to participate, they will be assigned to one of two groups which will receive different amounts of vitamin D. Subjects will be asked to keep a medication diary. Subjects may remain on treatment for approximately 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be greater than or equal to 18 years of age.
* Patients must have a newly diagnosed invasive ductal breast carcinoma, Stage I-II.
* Patients who have completed their surgical and radiation therapy.
* Patients must have SWOG performance status of 0, 1 or 2.
* Patients must have adequate organ function as defined by:
* Hgb > 8.0 gm/dl, WBC > 3,500, platelet count > 100,000
* Bilirubin < 2.0 mg/dl, SGOT < 4x upper limit of normal
* Creatinine < 2.0 mg/dl or calculated creatinine clearance > 50 ml/min
* Patients must have a serum calcium - phosphate product that is less than 70.
* Patients must have recovered from any prior surgery.
* Patients must be willing to use appropriate contraception if of child-bearing potential.
* Patients may be on standard of care maintenance dose Vit D3

Exclusion Criteria:

* Patients with histology of lobular carcinoma.
* Patients with metastatic disease.
* Pregnant or lactating women.
* Male gender.
* Patients with a history of sarcoidosis.
* Patients with any history of idiopathic urinary calcium stone disease, chronic hypercalcemia, or gastrointestinal malabsorptive conditions.
* Patients who have received any of the following treatments within the last 14 days prior to study registration will be excluded.
* Lithium
* Digitalis
* Thiazide diuretics
* Calcium supplementation during 1,25-dihydroxyvitamin D3 treatment
* Bisphosphonates
* Teriparatide
* Aluminum Hydroxide
* Bile Acid sequestrants
* Repletion dose VitD3 in setting of known Vit D3 deficiency or insufficiency
* Patients who have received concurrent corticosteroid treatments within the last 14 days prior to study registration will be excluded.
* Known HIV positive.
* Patients with an active infection requiring antibiotic therapy.
* Other malignancies unless the patient is considered to be disease-free for 5 or more years prior to randomization and is deemed by her physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Patients undergoing neoadjuvant chemotherapy or neoadjuvant endocrine therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Compare the differences in the T cell phenotype and function using PBMCs from patients in different cohorts | Prior to Treatment (Baseline), Week 4 and Week 8
  T cell analysis for the following markers will be evaluated-
  1. memory markers
  2. activation status and presence of regulatory T cells
  3. lymphoid organ-homing receptors
  4. Functional status of gated T cells will be analyzed
  5. cell surface thiol molecules and intracellular glutathione using flow cytometry to evaluate if anti-oxidant stus of the T cells is modulated in presence of the Vitamin D.
  These markers will help in determining the immunomodulatory potential of Vitamin D on T cell with respect to function, activation status and anti-oxidant capacity that can effect persistence and in turn immune outcome. The data obtained will be reported in terms of percent increase or decrease in number of T cells expressing particular receptors (homing or chemokine) or for differences in functional outcome (cytokine response) upon activation relative to samples collected at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States